CLINICAL TRIAL: NCT05134662
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled, Parallel Group Study to Evaluate the Safety and Tolerability, Pharmacodynamics and Pharmacokinetics of ALT-801 in Overweight and Obese Subjects With Type 2 Diabetes Mellitus
Brief Title: ALT-801 in Overweight and Obese Subjects With Type 2 Diabetes Mellitus (T2DM)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Altimmune, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ALT-801-104
Record Dates: First submitted 2021-11-15; First posted 2021-11-26 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Type 2 Diabetes
Keywords: Obese; Overweight; T2DM
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity; Overweight | interventions — ALT-801

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- ALT-801 1.2 mg (Experimental): 1.2 mg once weekly for 12 weeks
  Interventions: Drug: ALT-801
- ALT-801 1.8 mg (Experimental): 1.8 mg once weekly for 12 weeks
  Interventions: Drug: ALT-801
- ALT-801 2.4 mg (Experimental): 0.6 mg at Week 1, 1.2 mg at Week 2, 1.8 mg once weekly for 2 weeks (Weeks 3 and 4), and 2.4 mg once weekly for Weeks 5 through 12
  Interventions: Drug: ALT-801
- Placebo (Placebo Comparator): placebo once weekly for 12 weeks
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: ALT-801 — Injected subcutaneously (SC)
  Arms: ALT-801 1.2 mg; ALT-801 1.8 mg; ALT-801 2.4 mg
Other: Placebo — Injected subcutaneously (SC)
  Arms: Placebo

SUMMARY:
This is a Phase 1, randomized, double-blind, placebo-controlled, parallel group study to evaluate the safety and tolerability, pharmacodynamics (PD) and pharmacokinetics (PK) of ALT-801 and its effects on glucose control in overweight and obese subjects with type 2 diabetes mellitus (T2DM).

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent signed prior to the performance of any study procedures
* Male or female volunteers, age 18 to 65 years, inclusive
* Overweight to obese (BMI >/=28.0 kg/m2)
* Type 2 diabetes mellitus (T2DM), on stable regimen, for at least 3 months prior to screening, of any combination of (1) diet and exercise, (2) metformin with absent or mild gastrointestinal symptoms (nausea, vomiting or diarrhea), and/or (3) sodium glucose cotransporter-2 (SGLT-2) therapy
* Female subjects of childbearing potential who are not pregnant or breastfeeding, do not plan to become pregnant during the study, and agree to use effective birth control

Exclusion Criteria:

* Type 1 diabetes mellitus (DM) and/or insulin-dependent T2DM, or uncontrolled T2DM defined as hemoglobin A1c (HbA1c) ≥ 9.5% or C-peptide ≤ 8 ng/mL
* History of acute or chronic pancreatitis or hypersensitivity reaction to GLP-1 analogues

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2023-02-03 (Actual); Study Completion 2023-03-09 (Actual)

PRIMARY OUTCOMES:
The Number of Participants with One or More Treatment-Emergent Adverse Events (TEAEs) | Up to Day 110
Changes from baseline in area under the curve of serum glucose, C-peptide, and insulin | Baseline to Day 85
Changes from baseline in fasting serum glucose and insulin as measured by Homeostasis Model Assessment for Insulin Resistance 2 (HOMA-IR2) | Baseline to Day 85

SECONDARY OUTCOMES:
Change from baseline in fasting serum glucose | Baseline to Day 85
Change from baseline in hemoglobin A1c (HbA1c) | Baseline to Day 85

OTHER OUTCOMES:
Changes in quality of life questionnaires compared to baseline | Baseline to Day 85
ALT-801 concentrations | Baseline to Day 110
Change from baseline metformin concentrations | Baseline to Day 85

CONTACTS AND LOCATIONS:
Overall Officials: M. Scott Harris, MD, Study Director — Altimmune, Inc.
Locations (7):
- United States (7):
  - Altimmune CTM, Fort Myers, Florida
  - Altimmune CTM, Sarasota, Florida
  - Altimmune CTM, River Forest, Illinois
  - Altimmune CTM, Kansas City, Missouri
  - Altimmune CTM, Knoxville, Tennessee
  - Altimmune CTM, San Antonio, Texas
  - Altimmune CTM, Tomball, Texas